CLINICAL TRIAL: NCT05888259
Title: Changes in Plantar Pressure Distribution After 12 Weeks of Foot Insole Utility in Diabetic Foot Ulcer Patients: a Prospective, Randomized, Double-blinded, Controlled Clinical Trial
Brief Title: Plantar Pressure Distribution in Diabetic Foot Ulcer
Acronym: PPDDFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.P.T2207014
Record Dates: First submitted 2023-02-08; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot insole, medication and wound care (study group) (Experimental): Pressure maps were recorded to calculate peak pressures and pressure-time integrals for (hindfoot, middle foot, hallux, medial forefoot, and lateral forefoot).
  The measurements were uploaded to a server of software that uses technology to create a 3D model of the foot insole from multiple images taken by the user.
  Interventions: Other: foot insole
- medication and wound care (control group) (Active Comparator): participants will receive only medical treatments and wound care for the diabetic foot ulcer
  Interventions: Other: foot insole

INTERVENTIONS:
Other: foot insole — The foot insole is 5 mm thick under the flat part of the forefoot and the modification is done by changing the position of the metatarsal bar. This was another 5 mm above the flat part of the foot insole. The proximal/distal position of the metatarsal rod and the cavity distal to the rod (large cavity) were defined using the plantar pressure distribution. The position and shape of the distal end of the metatarsal bar were defined by a line in the area where the plantar pressure was 75% of the maximum plantar pressure The void measured 3 mm in depth.

SUMMARY:
The goal of this clinical trial is to find out the changes in peak pressure and pressure-time integral after twelve weeks from the initial utility of foot insoles and eight weeks later as a follow-up in diabetic foot ulcers. Participants will be randomly assigned to foot insole, medication, and wound care (study group) or medication and wound care (control group).

DETAILED DESCRIPTION:
Insole design The foot insole is 5 mm thick under the flat part of the forefoot and the modification is done by changing the position of the metatarsal bar. This was another 5 mm above the flat part of the foot insole. The proximal/distal position of the metatarsal rod and the cavity distal to the rod (large cavity) were defined using the plantar pressure distribution. The position and shape of the distal end of the metatarsal bar were defined by a line in the area where the plantar pressure was 75% of the maximum plantar pressure. This line also defined the void's proximal border. The void's distal border was housed near the area of peak plantar pressures, where pressure was 10% of peak plantar pressure. The void measured 3 mm in depth. After completing the initial design of the metatarsal bars and void, two variations were created by relocating the metatarsal bar proximal and distal by 2-4% of the insole length depending on the position of the foot ulcer. Based on a previous pilot study, this proportion equates to a distance of 5-7 mm on a size 38 orthotic insole. The orthotic insoles were made of medium-density (Ethylene-vinyl acetate) EVA (50° Shore A) and were manufactured on a CNC machine.

ELIGIBILITY:
* being between the ages of 50 and 65 years
* males and females
* with midfoot ulcer grades II or III
* diabetic foot ulcer
* the duration between 6 months and one year
* diabetes mellitus incidence between seven and ten years
* glycated hemoglobin between seven and nine (7 to 9%)
* body mass index between 25 and 30 kg|m2

Exclusion Criteria:

* Reynaud's disease
* peripheral arterial disease
* foot deformities
* foot burns.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
peak pressures | 12 weeks
  peak pressure for hindfoot, midfoot, hallux, medial and lateral forefoot
pressure-time integrals | 12 weeks
  pressure time integral for hindfoot, midfoot, hallux, medial, and lateral forefoot

CONTACTS AND LOCATIONS:
Overall Officials: Ebtsam H Allam, PHD, Principal Investigator — Cairo University; Hany M Elgohary, PHD, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elgohary HM, Al Jaouni SK, Selim SA. Effect of ultrasound-enhanced Nigella sativa seeds oil on wound healing: An animal model. J Taibah Univ Med Sci. 2018 Jun 27;13(5):438-443. doi: 10.1016/j.jtumed.2018.02.008. eCollection 2018 Oct. PMID 31435359